CLINICAL TRIAL: NCT06497712
Title: BEnefit of HYpnosis on Pain During Stitches in Emergency Room: the BE-HYPER Study
Brief Title: BEnefit of HYpnosis on Pain During Stitches in Emergency Room
Acronym: BE-HYPER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RBHP 2023 BOUILLON-MINOIS
Record Dates: First submitted 2024-05-29; First posted 2024-07-12 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Wound of Skin
Keywords: hypnosis; wound; stitches; pain; sinusal variability of cardiac frequency
MeSH Terms: conditions — Wounds and Injuries; Pain | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypnosis (Experimental): Patients will be hypnotized by a trained person before suturing.
  Interventions: Other: Hypnosis
- Standard of Care (No Intervention): Stitches will be performed without hypnosis as usual

INTERVENTIONS:
Other: Hypnosis — Before the beginning of stitches, the patient will be offered a hypnotic induction. The hypnotic induction is the initial phase of the hypnosis process. Its goal is to bring the patient to a state of dissociation: the hypnotic trance. Induction is usually achieved through progressive relaxation, sensory focusing, and a process of confusion.
  Arms: Hypnosis

SUMMARY:
Suturing is a daily practice in the emergency department, but it can be painful and stressful for patients. Hypnosis is increasingly used as a complement to the usual painkillers. The aim of our study was to investigate the impact of hypnosis on stitch placement in emergency department patients presenting with lacerations assessed by heart rate variability.

DETAILED DESCRIPTION:
The aim of this randomized, controlled, single-center, prospective study is to evaluate the impact of hypnosis during suturing in emergency department patients presenting with a laceration assessed by heart rate variability.

All patients with eligibility criteria will be included if the patient gave his written consent.

Patients will be randomized to one of two arms: (1) Hypnosis or (2) Standard Of Care (SOC) A heart rate monitoring belt will be fitted to the patient for both groups. The patient will be asked to complete a self-assessment questionnaire on pain and stress, as well as socio-demographic parameters.

A blood sample will be collected and the heart rate and blood pressure will be measured.

Stitches will be taken with or without hypnosis, and after 30 minutes, the pain and stress self-assessment questionnaire will again be completed by the patient, and a new blood test will be taken.

the heart rate monitoring belt will be removed, and the study will be completed for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years, admitted in Clermont-Ferrand University Hospital Emergency Department
* suturable wound
* patient's consent obtained

Exclusion Criteria:

* Pregnant or breast-feeding women
* Patient under guardianship, curators or safeguard of justice
* Person unable to give consent
* History of cardiac rhythm disorders (fibrillation, pacemaker)
* Psychiatric pathology
* Age < 18 years
* Surgical wound
* Eyelid, nose, ear or mouth wounds
* Patients who do not speak French
* Deaf patients
* Patients with no social security coverage
* Use of MEOPA
* Intake of toxic substances
* Head trauma with a Glasgow Score < or = to 14
* Patient with endocrinal pathologies on cortisol axe
* Refusal to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Impact of hypnosis during stitches among emergency department patients | Hour 0
  Impact of hypnosis will be evaluated by the variability of heart frequency measured by heart rate monitoring belt

SECONDARY OUTCOMES:
Impact of hypnosis on stress patients during stitches | Hour 0; Hour 0+30 minutes
  Visual analog scale (VAS) of pain and stress will be performed at two different times by the patient.
  A VAS is a 100-mm long horizontal line with verbal descriptors at each end to express the extremes of the feeling. Patients mark the point on the line that best corresponds to their pain and severity between 0 (no symptoms) to 100 (the worst pain and stress).
  Cut points on the pain VAS : no pain or low pain (0-29 mm), moderate pain (30-59 mm), and severe pain (>59 mm).
  Cut points on the stress VAS : no pain or low stress (0-19 mm), moderate stress (19-49 mm), severe stress (50-81 mm), and at-risk stress (>81 mm).
Evaluation of stress biomarkers in blood samples | Hour 0; Hour 0+30 minutes
  Evaluation of cortisol, DHEA, DHEA-s, ghrelin, leptin, IL-8, TNF-alpha, epinephrin, noradrenalin, dopamine
Evaluation of blood pressure | Hour 0; Hour 0+30 minutes
  Evaluation of hypnosis impact on systolic and diastolic blood pressure in millimeter of mercury (mmHg)
Evaluation of heart rate | Hour 0; Hour 0+30 minutes
  Evaluation of hypnosis impact on physiological parameters heart rate in beats per minute (bpm)
Impact of sociodemographics parameters on pain and stress | Hour 0; Hour 0+30 minutes
  Evaluation of the impact of sociodemographics parameters on pain and stress evaluated by the visual analog scale (VAS) performed at two different times (outcome N°2)
Impact of location of the wound on pain and stress | Hour 0; Hour 0+30 minutes
  Evaluation of the impact of location of the wound on stress and pain evaluated by the visual analog scale (outcome n°2)
Impact of location of the wound on variability of heart frequency | Hour 0; Hour 0+30 minutes
  Evaluation of the impact of location of the wound on the variability of heart frequency measured by heart rate monitoring belt (outcome n°1)
Impact of the length of the wound on pain and stress | Hour 0; Hour 0+30 minutes
  Evaluation of the impact of the length of the wound on stress and pain evaluated by the visual analog scale (outcome n°2)
Impact of the length of the wound on variability of heart frequency | Hour 0; Hour 0+30 minutes
  Evaluation of the impact of the length of the wound on the variability of heart frequency measured by heart rate monitoring belt (outcome n°1)
Impact of the depth of the wound on pain and stress | Hour 0; Hour 0+30 minutes
  Evaluation of the impact of the depth of the wound on stress and pain evaluated by the visual analog scale (outcome n°2)
Impact of the depth of the wound on pain and stress | Hour 0; Hour 0+30 minutes
  Evaluation of the impact of the depth of the wound on the variability of heart frequency measured by heart rate monitoring belt (outcome n°1)
sinusal variability of cardiac frequency on healthcare professional during stitching | Hour 0 and for 48 hours
  measurement of sinus variability of heart rate in healthcare professionals performing wound care by a heart rate transmitter holter positionned on the chest

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste BOUILLON-MINOIS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France